CLINICAL TRIAL: NCT02497417
Title: A Multi-Site Clinical Evaluation of the ARIES Clostridium Difficile Assay in Symptomatic Patients
Status: Completed | Type: Observational
Sponsor: Luminex Corporation (Industry)
Responsible Party: Sponsor
Organization: Luminex Molecular Diagnostics (Industry)
Other Study IDs: LMA-CDF-01-CS-001
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Gastroenteritis; Infectious Colitis
Keywords: ARIES Clostridium difficile
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool
Oversight: Data Monitoring Committee: No

SUMMARY:
The ARIES C. difficile Assay is a real-time PCR based qualitative in vitro diagnostic test for the direct detection of C. difficile nucleic acid in stool specimens.

DETAILED DESCRIPTION:
The ARIES C. difficile Assay is a real-time polymerase chain reaction (PCR) based qualitative in vitro diagnostic test for the direct detection of Clostridium difficile (C. difficile) nucleic acid in unformed (liquid or soft) stool specimens obtained from patients suspected of having Clostridium difficile associated disease (CDAD).

The objective of this study is to establish diagnostic accuracy of ARIES C. difficile Assay through a multi-site, method comparison on prospectively collected, left-over, stool specimens. Diagnostic accuracy will be expressed in terms of clinical sensitivity (or positive agreement) and specificity (or negative agreement).

ELIGIBILITY:
Inclusion Criteria:

* The specimen is from a patient suspected of having C. difficile associated disease (CDAD).
* The subject's specimen is an unpreserved, unformed (liquid or soft) stool submitted for testing at the site.

Exclusion Criteria:

* The specimen is preserved.
* The specimen was not properly collected, transported, processed or stored according to the instructions provided by the sponsor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All comers
Sampling Method: Probability Sample
Enrollment: 1021 (Actual)
Dates: Start 2016-10; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy will be a composite expressed in terms of clinical sensitivity (or positive agreement) and specificity (or negative agreement). | Within the first year of sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dunn, Study Director — Luminex Corporation
Locations (4):
- United States (4):
  - Tampa General Hospital, Tampa, Florida
  - Indiana University Health, Indianapolis, Indiana
  - TriCore Reference Laboratories, Albuquerque, New Mexico
  - The Ohio State University, Columbus, Ohio